CLINICAL TRIAL: NCT06871007
Title: Nivolumab and DA-EPOCH-R in Pediatric Primary Mediastinal (Thymic) Large B-cell Lymphoma
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director of RM Gorbacheva Research Institute, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 290
Record Dates: First submitted 2025-02-21; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Primary Mediastinal (Thymic) Large B-cell Lymphoma; Children; Nivolumab
MeSH Terms: interventions — Nivolumab; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisolone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The only ARM consists of nivolumab combined with DA-EPOCH-R protocol (Other): Children with PMLBL will receive standard chemotherapy (dose-adjusted EPOCH-R) combined with nivolumab 40 mg on Day 2
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 40 mg on Day 2 is added to dose-adjusted EPOCH-R (etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab; DA-EPOCH-R).Standard guidelines for conducting the DA-EPOCH-R protocol will be used.
  Other Names: Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisolone; Rituximab

SUMMARY:
Addition of nivolumab (immune checkpoint inhibitor) to standard chemotherapy (DA-EPOCH-R) may improve outcome in children with primary mediastinal large B-cell lymphoma

DETAILED DESCRIPTION:
A total of 6 blocks of Nivolumab+DA-EPOCH-R are planned for all patients regardless of stage and other risk factors. Nivolumab 40 mg (Day 2), Rituximab 375 mg/m2 (Day 1) and Prednisolone 60 mg/m2 (Days 1-5) are administered at constant unchangeable doses. Other drugs are administered at starting doses (Etoposide 50 mg/m2 (Days 1-4), Doxorubicin 10 mg/m2 (Days 1-4), Vincristine 0,4 mg/m2 (Days 1-4) and Cyclophosphamide 750 mg/m2 (Day 5). These starting doses are adjusted further according to standard principles of DA-EPOCH-R.

ELIGIBILITY:
Inclusion Criteria:

* Age from 0 years to 17 years 11 months

  * Established on the basis of histological and immunohistochemical studies, the diagnosis of PMLBL (the presence of programmed death-ligand on tumor cells is not necessary)
  * Lack of specific therapy for lymphoma
  * Signed informed consent

Exclusion Criteria:

* Age >18

  * History of specific therapy for lymphomas.
  * Drug intolerance

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 5 year
  Kaplan-Meyer estimate

SECONDARY OUTCOMES:
Overall survival | 5 year
  Kaplan-Meyer estimate
Progression free survival | 5 year
  Kaplan-Meyer estimate

CONTACTS AND LOCATIONS:
Overall Officials: Natalya Myakova, Principal Investigator — Dmitry Rogachev National Research Center; Ludmila Zubarovskaya, Principal Investigator — Pavlov University, R.M. Gorbacheva Research Institute
Locations (2):
- Russia (2):
  - Dmitry Rogachev National Research Center, Moscow
  - Pavlov University, RM Gorbacheva Research Institute, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No